CLINICAL TRIAL: NCT01216579
Title: Titrating Inhaled Steroid Dose Against Mannitol Hyper-responsiveness or BTS Outcomes: Comparative Effects on Asthma Exacerbations Over 1 Year
Brief Title: Steroid Titration Against Mannitol IN Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Professor Brian Jonathon Lipworth, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FARD002
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2008-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference arm (Placebo Comparator): Asthmatic patients managed as per British Thoracic Society guidelines by symptoms and lung function.
  Interventions: Other: mannitol (an airway challenge agent)
- Mannitol managed arm (Active Comparator): Group of asthmatic patients managed according to their mannitol challenge.
  Interventions: Other: mannitol (an airway challenge agent)

INTERVENTIONS:
Other: mannitol (an airway challenge agent)

SUMMARY:
The investigators hypothesise that titration of asthma medication against mannitol challenge results will reduce the number of mild asthma exacerbations, in one year, when compared with titration against BTS guidelines. To test this hypothesis the investigators propose a primary care, parallel treatment, patient blinded study in which matched groups of asthmatic patients will be treated in accordance either with BTS guidelines or with our treatment algorithm dependent on mannitol challenge result.

Purpose of the study is to evaluate the efficacy of a treatment algorithm based on the measurement of airway hyperresponsiveness to mannitol challenge, a surrogate marker of airway inflammation, in the long term treatment of asthma in comparison to BTS guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female asthmatics aged >/= 16 years
* Females must be non pregnant and non lactating
* FEV1 >/= 50% predicted
* Mannitol PD10 </= 635 mg at end of step down period
* No recent exacerbations of asthma requiring oral prednisolone in the previous 3 months
* Able to perform all the techniques necessary to carry out the challenge testing and lung function and compliant with taking the study medication
* Good inhaler technique which will be reinforced at each study visit

Exclusion Criteria:

* Male or female patients aged 15 or below
* FEV1 </= 50% predicted
* Patients who are currently taking a pulse of oral corticosteroids
* Patients with the following concomitant illnesses:bronchiectasis, allergic bronchopulmonary aspergillosis, COPD, heart failure, pulmonary fibrosis, rhino-sinusitis with polyps
* Immunocompromised patients
* Patients with recurrent LRTI
* Patients with documented aspirin induced asthma on LRTAs
* Pregnancy
* Known or suspected hypersensitivity to ICS or other excipients of the MDIs
* HIV/Hepatitis B or C positive

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2004-03; Primary Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lipworth, MD, Principal Investigator — University of Dundee

REFERENCES:
- [Derived] Anderson WJ, Short PM, Jabbal S, Lipworth BJ. Inhaled corticosteroid dose response in asthma: Should we measure inflammation? Ann Allergy Asthma Immunol. 2017 Feb;118(2):179-185. doi: 10.1016/j.anai.2016.11.018. Epub 2017 Jan 3. PMID 28065396
- [Derived] Anderson WJ, McFarlane LC, Lipworth BJ. Prospective follow-up of novel markers of bone turnover in persistent asthmatics exposed to low and high doses of inhaled ciclesonide over 12 months. J Clin Endocrinol Metab. 2012 Jun;97(6):1929-36. doi: 10.1210/jc.2011-3410. Epub 2012 Mar 21. PMID 22438232
- [Derived] Lipworth BJ, Short PM, Williamson PA, Clearie KL, Fardon TC, Jackson CM. A randomized primary care trial of steroid titration against mannitol in persistent asthma: STAMINA trial. Chest. 2012 Mar;141(3):607-615. doi: 10.1378/chest.11-1748. Epub 2011 Oct 13. PMID 21998259